CLINICAL TRIAL: NCT05784129
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of Guselkumab for the Treatment of Participants With Crohn's Disease After Surgical Resection
Brief Title: A Study of Guselkumab for the Treatment of Participants With Crohn's Disease After Surgical Resection
Acronym: PROGRESS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Janssen made an internal business decision to discontinue the PROGRESS study. This decision is not related to any efficacy or safety concerns.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109292; 2022-002389-33 (EudraCT Number); CNTO1959CRD3007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Crohn's Disease
Keywords: Endoscopy, Postoperative, Ileocolonic resection
MeSH Terms: conditions — Crohn Disease | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Guselkumab (Active Comparator): Participants will receive Guselkumab Dose 1 subcutaneously (SC) followed by Dose 2 SC thereafter through Week 144. Participants with disease recurrence will receive guselkumab SC treatment.
  Interventions: Drug: Guselkumab
- Group 2: Placebo (Placebo Comparator): Participants will receive matching placebo injections subcutaneously. Participants with disease recurrence will receive guselkumab SC treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered subcutaneously.
  Other Names: CNTO1959
  Arms: Group 1: Guselkumab
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of guselkumab treatment compared with placebo (an inactive substance with no medicine) in preventing recurrence of Crohn's disease in participants after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of Crohn's disease (CD) confirmed by endoscopic, histologic, and/or radiologic studies prior to resection or by tissue obtained at resection
* Have undergone an ileocolonic surgical resection (that is, an intestinal resection with an ileocolonic anastomosis) for CD prior to the baseline visit with the following criteria: (a)Have no known active CD anywhere in the gastrointestinal (GI) tract, including the findings at surgery. (b)Be able to undergo randomization no later than 49 days after surgery, and at least 10 days after surgery (or 8 days after resumption of bowel activity, example, in case of postoperative ileus) (c) Ileocolonic resection was not for the purpose of removing known dysplasia. (d) If ileocolonic resection is the participant's first resection for Crohn's, and occurs greater than (>) 10 years since the diagnosis of CD and only fibrostenotic stricturing is present, then length of stricture must be > 10 centimeter (cm)
* Have a baseline Crohn's Disease Activity Index (CDAI) less than (<) 200
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) test result during screening and a negative urine pregnancy test at week 0, prior to randomization
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 12 weeks after the last administration of study intervention

Exclusion Criteria:

* Has complications of CD, such as symptomatic strictures or stenoses, short bowel syndrome, a draining (that is, functioning) stoma or ostomy, or any other manifestation, that might be anticipated to require surgery, could preclude the use of the CDAI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with guselkumab
* Currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks before baseline, or 8 weeks before baseline for intra-abdominal abscesses, provided that there is no anticipated need for any further surgery
* Have had any active perianal disease within 3 months of screening (except skin tags) or have had any draining fistula within 3 months of screening unless the fistula was removed at the index surgery
* Evidence of a herpes zoster infection within 8 weeks before the first dose of study intervention
* Has a history of severe, progressive, or uncontrolled renal, genitourinary, hematologic, endocrine, cardiac, vascular, pulmonary, rheumatologic, neurologic, psychiatric, or metabolic disturbances, or signs and symptoms thereof

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- United States (9):
  - Medical Associates Research Group, Inc., San Diego, California
  - Gastroenterology Group Of Naples, Naples, Florida
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Gastro Health Ohio, Cincinnati, Ohio
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
- Poland (2):
  - Centrum Medyczne Medyk, Rzeszów
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4 participants who had recently undergone a surgical resection for Crohn's Disease (CD) were enrolled, randomized (1:1) and treated with study drug or placebo.
Pre-assignment Details: Due to early termination of the study, treatment period was up to Week 16 only. Participants were followed up for safety analysis till Week 28. The planned efficacy analysis was not performed due to the early study termination for reasons unrelated to safety or efficacy.
Groups:
- Guselkumab 200 mg + Guselkumab 100 mg: Participants were assigned to receive guselkumab 200 milligrams (mg) subcutaneous (SC) injection at Week 0 followed by guselkumab 100 mg SC injection at every 8 weeks thereafter until study termination (i.e., up to Week 16).
- Placebo: Participants were assigned to receive placebo matched to guselkumab SC injections at week 0 and at every 8 weeks thereafter until study termination (i.e., up to Week 16)
Period: Overall Study
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Started | 2 | 2
Treated at Weeks 0, 8 and 16 | 1 | 2
Treated at Weeks 0, 8 | 1 | 0
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Study terminated by sponsor | 2 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants. Based on the low enrolment number and in order to protect and maintain participant privacy/confidentiality, data were reported under a single arm.
Groups:
- Overall Participants: Participants received guselkumab 200 mg or matching placebo SC injection at Week 0 followed by guselkumab 100 mg or matching placebo SC injection at every 8 weeks thereafter until study termination (i.e., up to Week 16).
Arm/Group | Overall Participants
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (6.75)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 4
  From 65 to 84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic Recurrence Prior to or at Week 48
Description: Endoscopic recurrence was defined by modified Rutgeerts score greater than or equal to (>=) i2a in neo-terminal ileum, anastomotic site, or its equivalent in gastrointestinal (GI) tract (e.g., colonic ulceration). The modified Rutgeerts score ranged from i0 to i4, where i0 (No lesions), i1 (less than [<] 5 aphthous lesions), i2 (greater than [>] 5 aphthous lesions with normal mucosa between lesions or skip areas of larger lesions or lesions confined to ileocolonic anastomosis [<1 centimeter (cm) in length]), i2a (lesions confined to ileocolonic anastomosis [including anastomotic stenosis]), i2b (more than 5 aphthous ulcers or larger lesions, with normal mucosa in-between, in the neoterminal ileum [with or without anastomotic lesions]), i3 (diffuse aphthous ileitis with diffusely inflamed mucosa), i4 (large ulcers with diffuse mucosal inflammation or nodules or stenosis in neoterminal ileum). Higher score indicated worsening.
Time Frame: Baseline (Day 1) up to Week 48
Population: As no participant was available for the analysis due to early termination of study, no data was collected for this outcome measure.
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Clinical Remission Without Disease Recurrence at Week 48
Description: Clinical remission without disease recurrence at Week 48 was a composite endpoint defined by (1) Crohn's disease activity index (CDAI) <150 at Week 48 & (2) no endoscopic recurrence as defined by modified Rutgeerts score < i2a by Week 48 & (3) have not experienced disease recurrence. Disease recurrence was defined as (1) >=70 point increase from baseline in CDAI score at >8 weeks after randomization & CDAI score >=200 and evidence of endoscopic recurrence (Rutgeerts score <i2a) or (2) initiation of physician-prescribed corticosteroids or increase in steroid dose of >5 milligrams per day (mg/day) for treatment of Crohn's disease (CD) and endoscopic recurrence or (3) new draining or reopening of an internal or external fistula or (4) new perianal abscess or (5) new intra-abdominal abscess more than 3 months post index surgery. If a patient tested positive for enteric pathogen, infection should be treated and then participant should be reassessed for whether they meet disease recurrence.
Time Frame: At Week 48
Population: Due to early termination of the study, no formal data collection and analysis was possible and thus no data was collected for this outcome measure.
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Disease Recurrence
Description: Disease recurrence was defined by (1) a >=70 point increase from baseline in CDAI score at >8 weeks after randomization & CDAI score >=200 and evidence of endoscopic recurrence (Rutgeerts score <i2a) or (2) initiation of physician-prescribed corticosteroids or increase in steroid dose of >5 milligrams per day (mg/day) for treatment of Crohn's disease (CD) and endoscopic recurrence or (3) new draining or reopening of an internal or external fistula or (4) new perianal abscess or (5) new intra-abdominal abscess more than 3 months post index surgery. If a patient tested positive for enteric pathogen, infection should be treated and then participant should be reassessed for whether they meet disease recurrence.
Time Frame: Baseline (Day 1) up to Week 48
Population: as for outcome 2
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With No Abdominal Pain at Week 48
Description: Abdominal pain free at Week 48 is defined as abdominal pain (AP) score = 0 at Week 48. The scoring was done on a 4-point scale, ranged from 0 to 3, where 0 equals none, 1 equals mild, 2 equals moderate and 3 equals severe pain. Higher score indicated severe pain.
Time Frame: At Week 48
Population: as for outcome 2
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time To Recurrence of Symptoms
Description: Time-to-recurrence of symptoms was defined as time to attaining an AP mean daily score >1 (and also >1 point higher than baseline) along with stool frequency (SF) mean daily score >3 (and also >3 higher per day than baseline) for 2 consecutive weeks through Week 48. AP score scaling was done on a 4-point score scale, ranged from 0 to 3, where 0 equals none, 1 equals mild, 2 equals moderate and 3 equals severe pain. Higher score indicated severe pain. Stool frequency score was calculated from the total number of liquid or very soft stools in the previous 7 days.
Time Frame: Baseline (Day 1) up to Week 48
Population: as for outcome 2
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Number of participants with TEAEs and TESAEs were reported. An adverse event (AE) was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE/SAE occurring at or after the initial administration of study intervention through early termination of trial (up to Week 28) was considered to be treatment emergent.
Time Frame: Baseline (Day 1) up to early termination of trial (up to Week 28)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention and were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 2 | 2
Participants
  TEAEs | 1 | 1
  TESAEs | 1 | 1

7. Secondary Outcome: Serum Guselkumab Concentrations Over Time
Description: Serum guselkumab concentrations over time were reported. No summary analysis was done as study was terminated early and participant wise data were reported. This outcome measure was planned to be analyzed for "Guselkumab 200 mg + Guselkumab 100 mg" arm only.
Time Frame: At Weeks 0, 8, 16
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received at least 1 dose of study intervention, and had at least 1 valid blood sample drawn postbaseline for PK analysis and were analyzed according to the study intervention received. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number analyzed) signifies number of participants analyzed at specified categories.
Measure: Number; unit: micrograms/milliliters (ug/mL)
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg
Number analyzed (Participants) | 2
micrograms/milliliters (ug/mL)
  Participant 1 (Week 0): number analyzed (Participants) | 1
  Participant 1 (Week 0) | 0
  Participant 1 (Week 8): number analyzed (Participants) | 1
  Participant 1 (Week 8) | 1.68920
  Participant 1 (Week 16): number analyzed (Participants) | 1
  Participant 1 (Week 16) | 0.70957
  Participant 2 (Week 0): number analyzed (Participants) | 1
  Participant 2 (Week 0) | 0
  Participant 2 (Week 8): number analyzed (Participants) | 1
  Participant 2 (Week 8) | 2.87917

8. Secondary Outcome: Percentage of Participants With Steroid Free Clinical Remission at Week 48
Description: Steroid free clinical remission at Week 48 is defined as CDAI <150 and no corticosteroids within 30 days. The CDAI was a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. The CDAI score was assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s), and/or opiates, and general well-being. The last 4 variables were scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicated higher disease activities.
Time Frame: At Week 48
Population: as for outcome 2
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 12 weeks after last study dose administration (up to Week 28)
Description: Safety analysis set included all randomized participants who received at least 1 dose of study intervention and were analyzed according to the study intervention they actually received.
Arm/Group | Guselkumab 200 mg + Guselkumab 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guselkumab 200 mg + Guselkumab 100 mg (N=2) | Placebo (N=2)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early termination of study, protocol planned primary endpoint and few of secondary endpoints were not evaluable. Termination was not related to safety or efficacy of guselkumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT05784129/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05784129/SAP_001.pdf